CLINICAL TRIAL: NCT04880382
Title: Integrative Analysis of the Tumor Microenvironment and Optimization of the Immunotherapy Duration in Non-small Cell Lung Cancer Patients (OPTIMUNE-LUNG Study)
Brief Title: Integrative Analysis of Tumor Microenvironment and Optimization of Immunotherapy Duration in NSCL Cancer Patients
Acronym: OPTIMUNELUNG
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB 2019-07; 2020-005562-34 (EudraCT Number)
Record Dates: First submitted 2021-04-30; First posted 2021-05-10 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Immune checkpoint inhibition; non-small cell lung cancer; treatment duration; long-term benefit
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Randomized phase II study in which eligible patients will be randomized (1:1) according to two therapeutic strategies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Arm A: treatment by ICI will be continued (Other): After achieving objective response between 6 and 12 months after treatment onset, for these patients ICI treament will continue as per market authorization
  Interventions: Drug: ICI treatment continuation
- Experimental Arm B: treatment by ICI will be discontinued (Experimental): After achieving objective response between 6 and 12 months after treatment onset, for these patients first-line or second line regimen should be discontinued. Patients will be followed as per standard management.
  Interventions: Drug: ICI treatment discontinuation

INTERVENTIONS:
Drug: ICI treatment discontinuation — After achieving objective response between 6 and 12 months after treatment onset, for these patients, first or second line treatment by immune checkpoint inhibitor will be discontinued. Patients will be followed as per standard mangement thereafter
  Arms: Experimental Arm B: treatment by ICI will be discontinued
Drug: ICI treatment continuation — After achieving objective response between 6 and 12 months after treatment onset, for these patients, first or second line treatment by immune checkpoint inhibitor will be continued until disease progreession or unacceptable toxicity
  Arms: Standard Arm A: treatment by ICI will be continued

SUMMARY:
Non-comparative multicentric randomized study to assess long-term benefit of PD-1 inhibition in NSCLC patients who experienced a response between 6 and 12 months after initiation of ICI (immune checkpoint inhibitor PD1/PDL-1 blockade therapy)

DETAILED DESCRIPTION:
Two-arm, non-comparative, prospective, multicentric, randomized study for early discontinuation of immune checkpoint inhibitor PD1/PDL-1 blockade therapy in non-small cell lung cancer patients who achieved objective response between 6 and 12 months after treatment onset.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed non-small cell lung carcinoma (squamous or non squamous).
2. Locally advanced/unresectable or metastatic disease.
3. For non-squamous histology, tumor with no oncogenic addiction: no activating EGFR mutation, no ALK or ROS1 rearrangement,
4. Treatment with ICI (immune checkpoint inhibitor PD1/PDL-1 blockade therapy):

   1. in first or second-line treatment as per market authorization. For patients in first line, ICI alone or ICI + chemotherapy,
   2. start of ICI treatment 6 to 12 months (+/- 2 weeks) before registration.
5. At least one measurable lesion according to the RECIST v1.1 criteria before ICI treatment onset and confirmed by centralized review (lesion in previously irradiated filed can be considered as measurable if progressive at inclusion according to RECIST v1.1). At least one site of disease must be uni-dimensionally ≥ 10 mm.
6. Patient with objective response according to RECIST v1.1 criteria at 6 months or more and less than 12 months after ICI treatment onset. Response must be confirmed by centralized review
7. At least one lesion that can be biopsied for research purpose.
8. Age ≥ 18.
9. Performance status < 2.
10. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to registration.
11. Patient with a social security in compliance with the French law (Loi Jardé).
12. Patient must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
13. Voluntarily signed and dated written informed consent prior to any study specific procedure.

Exclusion Criteria:

1. Female who is pregnant or breast-feeding.
2. Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study.
3. Hypersensitivity to one of the active substances or to one of the excipients
4. Any contraindication to pursue ICI treatment as per investigator judgement.
5. Previous enrolment in the present study.
6. Individual deprived of liberty or placed under legal guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-08-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of the long-term benefit of PD-1 inhibition in NSCLC patients who experienced a response between 6 and 12 months after initiation of ICI | 12 months
  Long-term benefit will be assessed in terms of progression-free rate (PFR) at 12 months after randomization, for each therapeutic strategy

SECONDARY OUTCOMES:
Assessment of secondary resistance in NSCLC patients who experienced a response to PD1/PDL-1 inhibition | 12 months
  The rate of patients who develop progression (as per RECIST v1.1) due to secondary resistance after obtaining a response to PD1/PDL-1 inhibition, independently for each therapeutic strategy
Duration of response independently for each therapeutic strategy | Throughout the treatment period, an expected average of 12 months
  Duration of response (DoR) defined as the time interval between the first response (complete or partial response as per RECIST v1.1) to the time of the first documentation of disease progression
1-year progression-free survival, independently for each therapeutic strategy | 1 year
  Progression-free survival (PFS) defined as the time interval between the date of randomization and the date of progression or death, whichever occurs first. Progression will be determined according to RECIST v1.1
2-year progression-free survival, independently for each therapeutic strategy | 2 years
  Progression-free survival (PFS) defined as the time interval between the date of randomization and the date of progression or death, whichever occurs first. Progression will be determined according to RECIST v1.1
1-year overall survival, independently for each therapeutic strategy | 1 year
  Overall Survival (OS) defined as the time interval between the date of randomization and the date of death (of any cause)
2-year overall survival, independently for each therapeutic strategy | 2 years
  Overall Survival (OS) defined as the time interval between the date of randomization and the date of death (of any cause)
Safety profile, independently for each therapeutic strategy: Common Terminology Criteria for Adverse Events version 5 | Throughout the treatment and follow-up period, an expected average of 12 months
  Toxicity graded using the Common Terminology Criteria for Adverse Events version 5
• To describe retreatment for arm B-patients and subsequent systemic therapies for arm A-patients | Throughout the treatment and follow-up period, an expected average of 12 months
  Number of patients retreated by ICI will be described in Arm B. Similarly, for arm A-patients, number of patients treated by subsequent systemic therapy will be described
Tumor immune cells levels | At study onset (randomization) and at progression (throughout the treatment and follow-up period, an average of 12 months)
  Levels of immune cells in tumor will be measured by immunohistochemistry.
Blood cytokines levels | At study onset (randomization) and at progression (throughout the treatment and follow-up period, an average of 12 months)
  Levels of cytokines in blood will be measured by ELISA
Blood lymphocytes levels | At study onset (randomization) and at progression (throughout the treatment and follow-up period, an average of 12 months)
  Levels of lymphocytes in blood will be measured by flow cytometry
Blood kynurenine levels | At study onset (randomization) and at progression (throughout the treatment and follow-up period, an average of 12 months)
  Levels of kynurenine in blood will be measured by ELISA

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Centre Hospitalier de la Côte Basque, Bayonne
  - Clinique Tivoli Ducos, Bordeaux
  - Institut Bergonie, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Clinique Marzet, Pau

IPD SHARING:
Plan to Share IPD: No